CLINICAL TRIAL: NCT05945823
Title: A Phase 2 Study of Futibatinib in Combination With PD-1 Antibody-based Standard of Care Therapy in Patients With Solid Tumors.
Brief Title: Phase 2 Futibatinib in Combination With PD-1 Antibody Based Standard of Care in Solid Tumors
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Taiho Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAS-120-206
Expanded Access: NCT04507503 (Approved for marketing)
Record Dates: First submitted 2023-07-06; First posted 2023-07-14 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Locally Advanced Unresectable or Metastatic Solid Tumors Including Esophageal Cancer; Esophageal Adenocarcinoma; Esophageal Squamous Cell Cancer; Siewert Type 1 GEJ Cancer; Pancreatic Cancer
Keywords: Futibatinib; Advanced esophageal cancer; Esophageal cancer; TAS-120; Immunotherapy; Esophageal squamous cell cancer (ESCC); GEJ cancer; pancreatic ductal adenocarcinoma; pancreatic cancer
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma; Pancreatic Neoplasms; Esophageal Neoplasms | interventions — futibatinib; pembrolizumab; Cisplatin; Fluorouracil; Oxaliplatin; Leucovorin; Levoleucovorin; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): Patients with Esophageal cancer (Adenocarcinoma or Squamous cell cancer) will receive Futibatinib administered once daily on a continuous dosing regimen in combination with pembrolizumab plus investigator choice of SoC chemotherapy (FP or mFOLFOX6) for 6 cycles (induction phase) following by Futibatinib combination with pembrolizumab (consolidation phase).
  Interventions: Drug: Futibatinib; Drug: Pembrolizumab; Drug: Cisplatin; Drug: 5-FU; Drug: Oxaliplatin; Drug: Leucovorin; Drug: Levoleucovorin
- Cohort B (Experimental): Patients with PDAC will receive Futibatinib administered once daily on a continuous dosing regimen in combination with pembrolizumab plus mFOLFIRINOX for 6 cycles (induction phase) following by Futibatinib combination with pembrolizumab (consolidation phase) .
  Interventions: Drug: Futibatinib; Drug: Pembrolizumab; Drug: 5-FU; Drug: Oxaliplatin; Drug: Leucovorin; Drug: Levoleucovorin; Drug: Irinotecan

INTERVENTIONS:
Drug: Futibatinib — TAS-120 20 mg tablets, oral; once daily
  Other Names: TAS-120
Drug: Pembrolizumab — 400 mg once every 6-week-cycle, via IV infusion.
  Other Names: MK-3475; KEYTRUDA®
Drug: Cisplatin — 80 mg/m^2 Q3W via IV infusion, as part of investigator's choice FP chemotherapy
  Other Names: PLATINOL®
  Arms: Cohort A
Drug: 5-FU — 4000 mg/m^2 Q3W via IV infusion, as part of investigator's choice FP chemotherapy or 400 mg/m^2 Q2W via bolus IV infusion followed by 2400 mg/m^2 Q2W via continuous IV infusion, as part of investigator's choice mFOLFOX6 chemotherapy.
  2400 mg/m^2 Q2W via continuous IV infusion, as part of investigator's choice mFOLFOX6 chemotherapy.
  2400 mg/m^2 Q2W via continuous IV infusion, as part of mFOLFIRINOX chemotherapy.
  Other Names: ADRUCIL®
Drug: Oxaliplatin — 85 mg/m^2 Q2W via IV infusion, as part of mFOLFIRINOX or mFOLFOX6 chemotherapy. 2400 mg/m^2 Q2W via continuous IV infusion, as part of mFOLFIRINOX chemotherapy.
  Other Names: ELOXATIN®
Drug: Leucovorin — 400 mg/m^2 Q2W as part of mFOLFIRINOX or mFOLFOX6 chemotherapy.
  Other Names: calcium folinate; folinic acid; WELLCOVORIN®
Drug: Levoleucovorin — 200 mg/m^2 Q2W as part of investigator's choice mFOLFOX6 chemotherapy.
  Other Names: calcium levofolinate; levofolinic acid; FUSILEV®
Drug: Irinotecan — 150 mg/m^2 Q2W as part of mFOLFIRINOX chemotherapy.
  Arms: Cohort B

SUMMARY:
This is a nonrandomized, uncontrolled, open-label, multicenter Phase 2 study to evaluate the efficacy, safety, and tolerability of futibatinib in combination with PD-1 antibody-based SoC therapy in adult patients with solid tumors.

DETAILED DESCRIPTION:
Patients with locally advanced, unresectable or metastatic esophageal cancer (EC) or pancreatic ductal adenocarcinoma (PDAC) will receive futibatinib in combination with pembrolizumab plus standard of care (SOC) chemotherapy. Patients with EC will receive Investigator choice of chemotherapy (FP or mFOLFOX6), patients with PDAC will receive mFOLFIRINOX. Subjects will receive futibatinib in combination with pembrolizumab plus standard of care (SOC) chemotherapy during induction phase of the study and will continue on futibatinib in combination with pembrolizumab in consolidation phase.

ELIGIBILITY:
Inclusion criteria

1. Is ≥18 years of age at the time of informed consent
2. Cohort A: Histologically or cytologically confirmed, locally advanced, unresectable or metastatic adenocarcinoma or squamous cell carcinoma of the esophagus or advanced/metastatic Siewert type 1 adenocarcinoma of the esophagogastric junction (EGJ).
3. Cohort B: Histologically or cytologically confirmed, locally advanced, unresectable or metastatic pancreatic ductal adenocarcinoma.
4. No prior systemic treatment for locally advanced, unresectable or metastatic disease
5. Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) guidelines.
6. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
7. Adequate organ function
8. Able to take medications orally

Exclusion Criteria

1. Has locally advanced disease that is resectable or potentially curable with radiation therapy (as determined by local investigator).
2. Has an adenocarcinoma histology and is eligible to receive approved targeted therapy (eg, HER-2 positive patients).
3. Has received prior treatment with an anti-PD-1/PD-L1 or FGF/FGFR targeting drug, or any other agent directed to stimulatory or co-stimulatory T-cell receptor.
4. Has known additional malignancy that is progressing or requires active treatment.
5. History or current evidence of calcium and phosphate homeostasis disorder
6. Current evidence of clinically significant retinal disorder
7. Pregnant or lactating female.
8. Has known hypersensitivity or severe reaction to any of the study drugs or their excipients.
9. Has a diagnosis of immunodeficiency.
10. Has known human immunodeficiency virus (HIV) and/or history of Hepatitis B or C infections, or known to be positive for Hepatitis B antigen (HBsAg)/ Hepatitis B virus (HBV) DNA or Hepatitis C antibody or RNA.
11. Has an active autoimmune disease that has required systemic treatment in the past 2 years
12. Has a history of (noninfectious) pneumonitis that required steroids or has current pneumonitis.
13. Has had an allogenic tissue/organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2023-07-13 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
ORR by investigator assessment | 12 months
  Defined as the proportion of patients experiencing a best overall response of partial response (PR) or complete response (CR) (per RECIST 1.1), based on investigator assessment

SECONDARY OUTCOMES:
Treatment-emergent adverse events (TEAEs) as assessed by CTCAE v5.0 | 12 months
  Safety will be assessed based on reported AEs (including SAEs), graded by CTCAE V5.0., and dose modifications.
DoR per investigator assessment | 12 months
  defined as time from the first documentation of response to the first documentation of objective tumor progression or death due to any cause, whichever occurs first
DCR per investigator assessment | 12 months
  defined as percentage of patients who achieve complete response, partial response or stable disease per RECIST 1.1 by investigator assessment
PFS per investigator assessment | 12 months
  defined as the time from date of enrollment to the date of disease progression based on Investigator assessment of radiographic images or death, whichever occurs first
6-month PFS rate | 12 months
  defined as percentage of patients without disease progression within 6 months of enrollment

CONTACTS AND LOCATIONS:
Locations (22):
- United States (16):
  - University of California Los Angeles UCLA - Cancer Care - Santa Monica, Santa Monica, California
  - Rocky Mountain Cancer Centers Midtown, Denver, Colorado
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Henry Ford Health System, Detroit, Michigan
  - The Minniti Center - Medical Oncology and Hematology, Mickleton, New Jersey
  - Roswell Park Comprehensive Cancer Center (RPCCC) (Roswell Park Cancer Institute (RPCI)), Buffalo, New York
  - NYU Langone, New York, New York
  - Gabrail Cancer Center Research LLC, Canton, Ohio
  - Alliance Cancer Specialists, Horsham, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Dallas VA Medical Center, Dallas, Texas
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Blue Ridge Cancer Care, Roanoke, Virginia
  - Virginia Mason Medical Center, Seattle, Washington
  - Gundersen Lutheran Health System, La Crosse, Wisconsin
- France (2):
  - Centre Hospitalier Regional Universitaire de Lille, Lille
  - Centre Hospitalier Regional Universitaire Poitiers, Poitiers
- Germany (2):
  - Krankenhaus Nordwest gGmbH, Frankfurt
  - Universitaetsmedizin Mainz, Mainz
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid

IPD SHARING:
Plan to Share IPD: No